CLINICAL TRIAL: NCT06482294
Title: CIVETTA: Correlating Inflammatory Values of FEno, SympToms, SpuTum and Lung Function in Asthma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Alberto Papi, MD, professor, Università degli Studi di Ferrara
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 4739 - 2022-002677-29
Record Dates: First submitted 2024-06-25; First posted 2024-07-01 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Albuterol; Budesonide; Beclomethasone

STUDY DESIGN:
Intervention Model Description: crossover design according to the AB/BA scheme
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non ant-inflammatory rescue medication (Experimental): Salbutamol 200 mcg pMDI x2
  Interventions: Drug: Salbutamol
- Anti-inflammatory rescue medication (Experimental): (Salbutamol 200 mcg + either Fluticason 250 mcg DPI or Beclometasone 400 mcg DPI or Budesonide 400 mcg pMDI ) x2
  Interventions: Drug: Fluticason either Beclometasone or Budesonide

INTERVENTIONS:
Drug: Salbutamol — One arm is a combination of salbutamol and fluticason as a rescue medication (anti-inflammatory rescue medication). The second arm is salbutamol only as a rescue medication (non-anti-inflammatory rescue medication).
  Other Names: Salbutamol sulphate 200 mcg, pMDI
  Arms: Non ant-inflammatory rescue medication
Drug: Fluticason either Beclometasone or Budesonide — One arm is a combination of salbutamol and an ICS as a rescue medication (anti-inflammatory rescue medication). The second arm is salbutamol only as a rescue medication (non-anti-inflammatory rescue medication).
  Other Names: Fluticason Propionate 250 mcg DPI or Beclometasone dipropionate 400 mcg DPI or Budesonide 400 mcg pMDI or Budesonide 200 mcg DPI
  Arms: Anti-inflammatory rescue medication

SUMMARY:
Single-center, interventional, open-label, randomized phase II study aimed at describing the changes in airway inflammation at the onset of asthma symptoms that lead to the use of rapid acting bronchodilator (RABD) as a rescue medication in a mild to moderate asthma population. The study will assess whether there are differences in the airway inflammation profile in patients using a reliever medication containing ICS (anti-inflammatory rescue strategy) compared to a reliever medication containing only a bronchodilator for symptom relief (Non anti-inflammatory rescue strategy).

DETAILED DESCRIPTION:
The study is structured into two distinct and separate phases, an observational and an interventional.

- Phase 1: Observational Phase The observational component of the study aims to describe the variations in airway inflammation at the onset of asthma symptoms when patients (n=50) are under the appropriate anti-asthma therapy (Standard Of Care, SOC), which includes a rapid-onset bronchodilator (RABD) as needed. The RABD used may be either salbutamol or formoterol, depending on the therapeutic strategy employed by the patient and the GINA Track followed.

Before and after taking the SOC rescue medication, the patient will measure markers of airway inflammation and clinical impact (FeNO, FEV1, PEF, VAS scale) using the "PEFESP kit" provided to each enrolled patient. They will record these values in the "patient diary" for the subsequent 48 hours.

- Phase 2: Interventional Phase In a crossover design according to the AB/BA scheme, it will be assessed whether there are differences in the airway inflammation profile in patients (n=30) using a reliever medication containing ICS compared to a reliever medication containing only a bronchodilator.

The interventional phase consists of two open-label monitoring phases, each lasting a maximum of 3 weeks, separated by a washout period of 3 to 7 days and for a maximum of 3 symptom episodes. As in the observational part, patients will be asked to record the markers of airway inflammation and the clinical impact of symptoms at the onset of the change from stable condition and in the 48 hours following the administration of the reliever medication.

Patient with mild asthma will be the first group of severity enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients already followed for asthma according to ERS/ATS criteria
* Mild and moderate asthma (GINA steps 1-3), with the exclusion of patients with severe asthma (GINA steps 4-5).

Exclusion Criteria:

Severe asthma (Gina steps 4 and 5)

* Inability to give informed consent
* Diagnosis of other clinically significant respiratory diseases
* Diagnosis of Chronic Obstructive Pulmonary Disease (COPD)
* History of smoking: > 10 pack/year or stop for less than 3 months
* Oral steroid therapy in the 2 months prior to enrollment
* Number of asthma exacerbations per year ≥ 2
* Pregnancy
* Evidence of clinically significant pathologies other than in respiratory system (i.e., cardiovascular, hepatic, renal, nervous, endocrinological, oncological, dermatological systems)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate airway inflammation characteristics and changes at the onset of asthma symptoms requiring as-needed therapy (RABD) and the impact of inhaled steroid therapy in addition to RABD on airway inflammation | Patients are asked to perform repeated measurements of airway inflammation from the onset of symptoms to 48 hours after the administration of the rescue medication.
  Inflammation will be assessed as FeNO levels after an anti inflammatory rescue medication compared to a non anti inflammatory rescue medication therapy repeatedly measured up to 48 hours at defined intervals

SECONDARY OUTCOMES:
Change in FEV1 | Patients are asked to perform repeated measurements of FEV1 from the onset of symptoms to 48 hours after the administration of the rescue medication.
  The change in FEV after administration of an anti-inflammatory rescue medication and a non-anti-inflammatory rescue medication.
change in Visual Analogue Scale (VAS) scale. | Patients are asked to perform repeated measurements of VAS scale from the onset of symptoms to 48 hours after the administration of the rescue medication.
  The change in VAS scale, used to measure the intensity of symptoms (0 lowest intensity, 10 highest intensity) after administration of an anti-inflammatory rescue medication and a non-anti-inflammatory rescue medication.

OTHER OUTCOMES:
Change in sputum eosinophils count | Patients are asked to perform repeated sputum collections from the onset of symptoms until 48 hours after the administration of the rescue medication.
  The change in sputum eosinophils count after administration of an anti-inflammatory rescue medication and a non-anti-inflammatory rescue medication.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Papi, MD, Principal Investigator — Università degli Studi di Ferrara
Locations (1):
- Research Centre on Asthma and COPD, University of Ferrara, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: No